CLINICAL TRIAL: NCT07101133
Title: Research on Key Technologies of Precision Nutrition for Obesity Intervention
Brief Title: Precision Nutrition Technologies for Obesity Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuan He (Other)
Responsible Party: Sponsor-Investigator, Yuan He, Researcher, professor, doctoral supervisor,, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2023ZD0508300
Record Dates: First submitted 2025-06-09; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Obesity and Obesity-related Medical Conditions
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group: Energy-limited balanced diet group (Placebo Comparator): Standardized energy-restricted balanced dietary intervention was provided. The intake for men was 1350kcal/d, and for women it was 1100kcal/d. The proportions of the three major nutrients were 50-65% carbohydrates, 20-30% fats, and 15-20% proteins.
  Interventions: Dietary Supplement: Control group: Energy-limited balanced diet group
- Intervention group based on clinical phenotype (Experimental): Based on subjects baseline diet quality assessment (by FFQ questionnaires and 3 diet records) and baseline clinical data (blood glucose, blood lipid, CRP, etc.), formulate diet plan, targeted adjust the types and proportions of food, mainly includes the following three types: Scheme 1: A low fat diet intake of 1350 kcal/d pattern men, women of 1100 kcal/d, compared with three major nutrients carbohydrate 62%, fat 20%, protein 18%. Scheme 2: low carbohydrate diet intake of 1350 kcal/d pattern men, women of 1100 kcal/d, three major nutrients ratio of carbohydrate, 37% fat, 45% protein, 18%. Solution 3: limited energy balanced diet provide a standardized and balanced energy-restricted diet (1,350 kcal/d for men and 1,100 kcal/d for women), with the proportion of the three major nutrients being 54% carbohydrates, 28% fats, and 18% proteins. Staple meal replacement: Replace two meals a day with full-nutrition meal replacement , wwith a calorie content of 30 to 40%.
  Interventions: Dietary Supplement: Control group: Energy-limited balanced diet group
- Intervention group based on genetic susceptibility (Experimental): Integrate deep phenotypes (diet quality, physical fitness test results, clinical indicators), superimpose obesity nutrition gene data, including the test results of 33 obesity-related genes (such as FTO, MC4R) and nutrient metabolism genes (such as APOA2, PPARG), and customize the macronutrient ratio (such as adopting a low-carbohydrate diet for those with high carbohydrate sensitivity). Dietary patterns mainly include low-fat dietary patterns, low-carb and low-fat dietary patterns, and balanced energy-restricted dietary patterns. Staple meal replacement: The same meal replacement plan as the deep phenotype group.
  Interventions: Dietary Supplement: Control group: Energy-limited balanced diet group
- Based on genetic susceptibility + intestinal flora intervention group (Experimental): Integrating deep phenotypes (diet quality, physical fitness test results, clinical indicators), superimposing obesity nutrition gene + intestinal flora genomic data, including 33 obesity nutrition-related genes and 170 intestinal obesity nutrient metabolic bacterial genera/species test results, to customize the proportion of macronutrients. Dietary patterns mainly include low-fat dietary patterns, low-carb and low-fat dietary patterns, and balanced energy-restricted dietary patterns. Staple meal replacement: The same meal replacement plan as the deep phenotype group.
  Interventions: Dietary Supplement: Control group: Energy-limited balanced diet group

INTERVENTIONS:
Dietary Supplement: Control group: Energy-limited balanced diet group — Based on clinical phenotype + energy-restricted diet group：Based on the baseline dietary quality assessment of the subjects and baseline clinical data , a dietary plan was formulated, and the types and proportions of food were adjusted specifically .
  Intervention group based on genetic susceptibility：Integrate deep phenotypes (diet quality, physical fitness test results, clinical indicators), superimpose obesity nutrition gene data and nutrient metabolism genes, and customize the macronutrient ratio.
  Based on genetic susceptibility + intestinal flora intervention group: Integrating deep phenotypes (diet quality, physical fitness test results, clinical indicators), superimposing obesity nutrition gene + intestinal flora genomic data, including 33 obesity nutrition-related genes and 170 intestinal obesity nutrient metabolic bacterial genera/species test results, to customize the proportion of macronutrients.
  Other Names: Based on clinical phenotype + energy-restricted diet group; Intervention group based on genetic susceptibility; Based on genetic susceptibility + intestinal flora intervention group

SUMMARY:
The implementation of this project will develop and apply precision health dietary solutions tailored for weight management in China's obese population, establishing a precision nutrition intervention model. Over 50% of the obese individuals are expected to achieve a weight reduction of more than 5%, significantly improving their quality of life.

ELIGIBILITY:
Inclusion Criteria:18 years old to 60 years old, gender not limited. Obesity diagnosis standard, 28≤ BMI (kg/m2)≤ 35 ; Signed informed consent;

Exclusion Criteria:Secondary obesity caused by endocrine, genetic, central nervous system diseases or drugs; Merge major disease, tumor, each system organ failure; Had serious infection and acute cardiocerebrovascular diseases; Over the past three months in three months, or drug or surgical treatment has been put on a diet; Pregnancy, for pregnant and nursing women; Mental disorders, or physical/body movement disorders affect normal activities; 5 kg weight fluctuation in the past two months; Daily alcohol consumption quantity more than 25 g for man, women more than 15 g.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-07-27 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight and BMI ;Changes in abdominal fat (waist circumference, waist-to-height ratio, visceral fat area in the abdomen), and body fat percentage. | 3 months
  Individuals whose weight changes during the weight loss period exceed 5% of their own body weight; dropout rates during weight loss and maintenance periods

REFERENCES:
- [Background] Gong P, Liang S, Carlton EJ, Jiang Q, Wu J, Wang L, Remais JV. Urbanisation and health in China. Lancet. 2012 Mar 3;379(9818):843-52. doi: 10.1016/S0140-6736(11)61878-3. PMID 22386037
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Trends in adult body-mass index in 200 countries from 1975 to 2014: a pooled analysis of 1698 population-based measurement studies with 19.2 million participants. Lancet. 2016 Apr 2;387(10026):1377-1396. doi: 10.1016/S0140-6736(16)30054-X. PMID 27115820